CLINICAL TRIAL: NCT01595373
Title: Local Metabolic Effects of Ghrelin: A Clinical Microdialysis Study
Brief Title: Local Metabolic Effects of Ghrelin in Skeletal Muscle and Adipose Tissue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Esben Thyssen Vestergaard (Other)
Responsible Party: Sponsor-Investigator, Esben Thyssen Vestergaard, Postdoc PhD, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012-28512
Record Dates: First submitted 2012-05-07; First posted 2012-05-10 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Ghrelin; Microdialysis; Controls; Metabolic effects of ghrelin
MeSH Terms: interventions — acyl-ghrelin; Ghrelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ghrelin (Active Comparator): Ghrelin
  Interventions: Drug: Acyl ghrelin
- Placebo (Placebo Comparator): Ringer acetate is used for placebo.
  Interventions: Drug: Placebo (Ringer acetate)

INTERVENTIONS:
Drug: Acyl ghrelin — Acyl ghrelin 12.5 pg/min infused continuously for 300 minutes
  Other Names: Human acyl ghrelin; Ghrelin
  Arms: Ghrelin
Drug: Placebo (Ringer acetate) — Ringer acetate 2 microliter/min for 300 minutes
  Arms: Placebo

SUMMARY:
The metabolic effects of ghrelin is investigated by microdialysis technique. Subjects are healthy young men. End points are interstitial concentrations of glucose, lactate, and glycerol.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* age 18-65 years (included)
* Body mass index 20-25 (included)

Exclusion Criteria:

* alcohol abuse
* malignant disease
* use of any medicine except otc painkillers
* any disease recognized
* participation in a trial using radioactive isotopes within the last 6 months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Interstitial concentrations of glycerol | Interstitial concentrations of glycerol at t=120 minutes

SECONDARY OUTCOMES:
Interstitial concentrations of lactate | Interstitial concentrations of lactate at t=120 minutes
Interstitial concentrations of glucose | Interstitial concentrations of glucose at t=120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Esben T. Vestergaard, MD PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Vestergaard ET, Moller N, Jorgensen JO. Acute peripheral tissue effects of ghrelin on interstitial levels of glucose, glycerol, and lactate: a microdialysis study in healthy human subjects. Am J Physiol Endocrinol Metab. 2013 Jun 15;304(12):E1273-80. doi: 10.1152/ajpendo.00662.2012. Epub 2013 Apr 16. PMID 23592479